CLINICAL TRIAL: NCT00954356
Title: Single-Center, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Proof-of-Concept Study to Evaluate the Safety, PK, & Efficacy of a Single Oral Dose of XPF-001 in the Treatment of Pain Related to Third Molar/Wisdom Tooth Extraction.
Brief Title: Safety and Efficacy Study of XPF-001 to Treat Pain Following Wisdom Tooth Extraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XPF-001-201
Record Dates: First submitted 2009-07-22; First posted 2009-08-07 (Estimated); Results first posted 2012-06-29 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Dental Pain
Keywords: Pain following 3rd molar/wisdom tooth extraction
MeSH Terms: conditions — Toothache

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- XPF-001 (Experimental)
  Interventions: Drug: XPF-001
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: XPF-001 — Single oral administration of 500 mg XPF-001 capsules (5 x 100 mg capsules)
  Arms: XPF-001
Drug: placebo — Single oral administration of 5 x 100 mg Placebo capsules.
  Arms: Placebo

SUMMARY:
The purpose of this trial is to determine if XPF-001 is effective for the treatment of pain following third-molar/wisdom tooth extraction.

ELIGIBILITY:
Inclusion Criteria:

* Males (aged 18-60) and females of non-childbearing potential (aged 18-60;
* BMI between 19.5 to 32.0 kg/m2;
* Outpatient, scheduled to undergo surgical extraction of 2 or more impacted 3rd molars (with at least 1 partial bony mandibular extraction);
* use of only the following preoperative medications 2% lidocaine with epinephrine and nitrous oxide;
* Able to complete the requested information on analgesic questionnaires and able to comply with study procedures and restrictions;
* Able to read, comprehend and sign the consent form;
* Deemed medically healthy to participate in the study, with normal or clinically insignificant medical history, physical examination, lab tests and ECG results;
* No contraindications to the study drug, it excipients or any of the study medications including rescue medications.

Exclusion Criteria:

* Presence of a clinically significant medical condition;
* Positive test for HIV, Hepatitis B or Hepatitis C;
* Use of any prescription or over the counter medication or supplement in the 48 hours before dose of study drug until discharge;
* Acute local infection at the time of dental surgery;
* Females who are pregnant, lactating or of child-bearing potential, or who provide a positive pregnancy test result at screening or check-in;
* Males not undertaking adequate measures to prevent their partner becoming pregnant throughout the study;
* Clinically significant laboratory values;
* Clinically significant abnormal ECG;
* History or presence of alcoholism, or alcohol or substance abuse (within previous 2 years), or routine consumption of 3 or more alcoholic drinks per day;
* A positive urine drug test;
* Routine use of analgesics 5 or more times per week;
* Presence or history (within 2 years of enrolment) of bleeding disorder(s) or peptic ulcer disease;
* History of allergic reaction to any drug, including penicillin;
* Ingestion of caffeine containing foods or drinks in the 24 hours before dose of study drug;
* Consumption of alcohol in the 48 hours before dose of study drug, or a positive alcohol breath test at check-in;
* Consumption of grapefruit or grapefruit containing products in the 7 days before dose of study drug;
* Use of tobacco or nicotine substitutes within 1 month of dose of study drug, or inability to refrain from use of nicotine between check-in and follow up;
* Treatment for depression in the 6 months prior to enrolment;
* Use of another investigational drug in the 60 days before enrolment;
* Donation or loss of 50-500 mL of blood in the 30 days prior to enrolment, or more than 500 mL of blood in the 56 days before enrolment;
* Previously entered into this study;
* Study site or Sponsor employees or relatives of employees directly involved in the study;
* Any other condition that (in the opinion of the Investigator or sponsor) makes the subject unsuitable for the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Christensen, DDS, Principal Investigator — Jean Brown Research
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All 61 subjects were recruited at a single center between September 29th and November 16th 2009.
Groups:
- XPF-001: 500 mg XEN402 (5x 100 mg capsules) administered as a single dose
- Placebo: 5 x matching placebo capsules (administered as a single dose)
Period: Overall Study
Arm/Group | XPF-001 | Placebo
Started | 41 | 20
Completed | 41 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XPF-001 | Placebo | Total
Number analyzed (Participants) | 41 | 20 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 20 | 61
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 20.2 (2.94) | 20.9 (3.01) | 20.4 (2.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 41 | 20 | 61
Region of Enrollment [Number; unit: participants]
  United States | 41 | 20 | 61

OUTCOME MEASURES:

1. Primary Outcome: Total Pain Relief at 6 Hours Post Dose (TOTPAR 6)
Description: The primary efficacy variable was total pain relief at the 6-hour observation (TOTPAR 6); TOTPAR 6 is an area calculation incorporating time and relief scores over the 6 hours following dosing and was calculated using Simpson's trapezoidal rule.
  The higher the LS Means scores, the more pain relief was obtained.
  Relief (REL) scores were measured at multiple timepoints after dosing, using a 5 point categorical pain relief rating scale. (None = 0, A Little Relief = 1, Some = 2, A Lot = 3, Complete Relief = 4). The minimum possible TOTPAR 6 score = 0, maximum possible score = 24
Time Frame: 6 hours post dose
Population: Published data from an impacted wisdom tooth removal was used to determine a 60 subject study with 2:1 randomisation and a one-sided significance level of 0.10 would have a power of 84.1%. LOCF was used for imputed values and all subjects were included in both the IIT and PP populations for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Placebo: Subjects received a single dose of placebo after reaching moderate pain on a numerical rating scale following surgical extraction of 2 or more impacted third molars, of which at least 1 was a partial or full bony mandibular impaction.
- XPF-001: Subjects received a single dose of XPF-001 500 mg after reaching moderate pain on a numerical rating scale following surgical extraction of 2 or more impacted third molars, of which at least 1 was a partial or full bony mandibular impaction.
Arm/Group | Placebo | XPF-001
Number analyzed (Participants) | 20 | 41
units on a scale | 2.45 [0.182 to 4.72] | 4.37 [2.79 to 5.96]

2. Secondary Outcome: Total Pain Relief (TOTPAR) at 4 Hours Post Dose
Description: A secondary efficacy variable was total pain relief at the 4-hour observation (TOTPAR 4); TOTPAR 4 is an area calculation incorporating time and relief scores over the 4 hours following dosing and was calculated using Simpson's trapezoidal rule.
  The higher the LS Means scores, the more pain relief was obtained.
  Relief (REL) scores were measured at multiple timepoints after dosing, using a 5 point categorical pain relief rating scale. (None = 0, A Little Relief = 1, Some = 2, A Lot = 3, Complete Relief = 4). The minimum possible TOTPAR 4 score = 0, maximum possible score = 16).
Time Frame: 4 hours
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | XPF-001
Number analyzed (Participants) | 20 | 41
units on a scale | 1.51 [0.214 to 2.81] | 2.44 [1.54 to 3.35]

3. Secondary Outcome: Total Pain Relief (TOTPAR) at 8 Hours Post Dose
Description: A secondary efficacy variable was total pain relief at the 8-hour observation (TOTPAR 8); TOTPAR 8 is an area calculation incorporating time and relief scores over the 8 hours following dosing and was calculated using Simpson's trapezoidal rule.
  The higher the LS Means scores, the more pain relief was obtained.
  Relief (REL) scores were measured at multiple timepoints after dosing, using a 5 point categorical pain relief rating scale. (None = 0, A Little Relief = 1, Some = 2, A Lot = 3, Complete Relief = 4). The minimum possible TOTPAR 8 score = 0, maximum possible score = 32
Time Frame: 8 hours
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | XPF-001
Number analyzed (Participants) | 20 | 41
units on a scale | 3.43 [0.126 to 6.73] | 6.41 [4.11 to 8.71]

4. Secondary Outcome: Total Pain Relief (TOTPAR) at 12 Hours Post Dose
Description: A secondary efficacy variable was total pain relief at the 12-hour observation (TOTPAR 12); TOTPAR 12 is an area calculation incorporating time and relief scores over the 12 hours following dosing and was calculated using Simpson's trapezoidal rule.
  The higher the LS Means scores, the more pain relief was obtained.
  Relief (REL) scores were measured at multiple timepoints after dosing, using a 5 point categorical pain relief rating scale. (None = 0, A Little Relief = 1, Some = 2, A Lot = 3, Complete Relief = 4). The minimum possible TOTPAR 12 score = 0, maximum possible score = 48.
Time Frame: 12 hours
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | XPF-001
Number analyzed (Participants) | 20 | 41
units on a scale | 5.42 [-0.019 to 10.9] | 10.7 [6.93 to 14.5]

5. Secondary Outcome: Summed Pain Intensity Difference (SPID) at 4 Hours Post Dose
Description: Pain intensity was scored on an 11-point scale (PINRS), (0=no pain - 10=pain as bad as you can imagine). Scores were measured at baseline (after surgery but before dosing) and at multiple timepoints after dosing. At each timepoint, pain intensity difference (PID) was calculated (ie, baseline score minus timepoint score).
  SPID4 is an area calculation encompassing time and the PID scores over the 4 hours following dosing. The minimum possible SPID4 value = -40, the maximum possible = 40.
  A positive SPID LS Means score implies reduced pain intensity over the corresponding time period.
Time Frame: Baseline to 4 hours post dose
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | XPF-001
Number analyzed (Participants) | 20 | 41
units on a scale | -0.577 [-3.55 to 2.39] | 0.364 [-1.71 to 2.43]

6. Secondary Outcome: Summed Pain Intensity Difference (SPID) at 6 Hours Post Dose
Description: Pain intensity was scored on an 11-point scale (PINRS), (0=no pain - 10=pain as bad as you can imagine). Scores were measured at baseline (after surgery but before dosing) and at multiple timepoints after dosing. At each timepoint, pain intensity difference (PID) was calculated (ie, baseline score minus timepoint score).
  SPID6 is an area calculation encompassing time and the PID scores over the 6 hours following dosing. The minimum possible SPID6 value = -60, the maximum possible = 60.
  A positive SPID LS Means score implies reduced pain intensity over the corresponding time period.
Time Frame: Baseline to 6 hours post dose
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | XPF-001
Number analyzed (Participants) | 20 | 41
units on a scale | -0.811 [-5.89 to 4.26] | 1.48 [-2.06 to 5.02]

7. Secondary Outcome: Summed Pain Intensity Difference (SPID) at 8 Hours Post Dose
Description: Pain intensity was scored on an 11-point scale (PINRS), (0=no pain - 10=pain as bad as you can imagine). Scores were measured at baseline (after surgery but before dosing) and at multiple timepoints after dosing. At each timepoint, pain intensity difference (PID) was calculated (ie, baseline score minus timepoint score).
  SPID8 is an area calculation encompassing time and the PID scores over the 8 hours following dosing. The minimum possible SPID8 value = -80, the maximum possible = 80.
  A positive SPID LS Means score implies reduced pain intensity over the corresponding time period.
Time Frame: Baseline to 8 hours post dose
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | XPF-001
Number analyzed (Participants) | 20 | 41
units on a scale | -0.958 [-8.24 to 6.33] | 2.77 [-2.31 to 7.85]

8. Secondary Outcome: Summed Pain Intensity Difference (SPID) at 12 Hours Post Dose
Description: Pain intensity was scored on an 11-point scale (PINRS), (0=no pain - 10=pain as bad as you can imagine). Scores were measured at baseline (after surgery but before dosing) and at multiple timepoints after dosing. At each timepoint, pain intensity difference (PID) was calculated (ie, baseline score minus timepoint score).
  SPID12 is an area calculation encompassing time and the PID scores over the 12 hours following dosing. The minimum possible SPID12 value = -120, the maximum possible = 120.
  A positive SPID LS Means score implies reduced pain intensity over the corresponding time period.
Time Frame: Baseline to 12 hours post dose
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | XPF-001
Number analyzed (Participants) | 20 | 41
units on a scale | -1.10 [-13.0 to 10.8] | 5.68 [-2.60 to 14.0]

9. Secondary Outcome: Time to First Perceptible Relief
Description: Onset of analgesia was measured using 2 stopwatches. Both stopwatches were started at the time of dose administration. Stopwatch 1 was pressed by the subject when any pain relief was first perceived (Time to First Perceptible Relief) and stopwatch 2 was pressed by the subject when pain relief became meaningful (Time to Meaningful Relief).
Time Frame: 24 hours
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | XPF-001
Number analyzed (Participants) | 20 | 41
Minutes | NA [37 to NA] — Data not estimable as less than 50% of subject reported perceptible relief. A minimum of 50% of subjects are required to report the event in order to calculate the median. | NA [59 to NA] — Data not estimable as less than 50% of subject reported perceptible relief. A minimum of 50% of subjects are required to report the event in order to calculate the median.

10. Secondary Outcome: Time to Meaningful Relief
Description: Onset of analgesia was measured using 2 stopwatches. Both stopwatches were started at the time of dose administration. Stopwatch 1 was pressed by the subject when any pain relief was first perceived (Time to First Perceptible Relief) and stopwatch 2 was pressed by the subject when pain relief became meaningful (Time to Meaningful Relief).
  'Meaningful Relief' was defined as when the relief became 'meaningful' to each individual subject, and was not necessarily a complete absence of pain. 'Meaningful Relief' could not occur before 'First Perceptible Relief'.
Time Frame: 24 hours
Measure: Median (90% Confidence Interval); unit: Minutes
Arm/Group | Placebo | XPF-001
Number analyzed (Participants) | 20 | 41
Minutes | NA [NA to NA] — Data not estimable as less than 50% of subject reported meaningful relief. A minimum of 50% of subjects are required to report the event in order to calculate the median. | NA [NA to NA] — Data not estimable as less than 50% of subject reported meaningful relief. A minimum of 50% of subjects are required to report the event in order to calculate the median.

11. Secondary Outcome: Time to Rescue Medication
Description: The time of administration of rescue medication (if any) was recorded for each subject and the duration since dosing was calculated.
Time Frame: 24 hours
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | XPF-001
Number analyzed (Participants) | 20 | 41
Minutes | 93 [73 to 153] | 133 [103 to NA] — The upper limit of the 95% confidence interval is not calculable from the available data.

12. Secondary Outcome: Treatment Emergent Adverse Events
Description: Adverse Events were recorded at the time of occurence. Clinically significant findings (if any) in ECG and vital signs assessments and laboratory samples were recorded as adverse events.
  Treatment Emergent Adverse Events (TEAEs) are those which either started or worsened following administration of study drug (XPF-001 or placebo).
Time Frame: 48 hours
Measure: Number; unit: Events
Arm/Group | Placebo | XPF-001
Number analyzed (Participants) | 20 | 41
Events | 7 | 35

ADVERSE EVENTS:
Arm/Group | XPF-001 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/20
Other Adverse Events (participants affected / at risk) | 16/41 | 4/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | XPF-001 (N=41) | Placebo (N=20)
Dizziness (Nervous system disorders) | 7 | 0
Somnolence (Nervous system disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 8 | 2
Neutrophil count increased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Confusional State (Psychiatric disorders) | 3 | 0
Headache (Nervous system disorders) | 4 | 1

LIMITATIONS AND CAVEATS:
This model is best suited for drugs with rapid onset of action (e.g. NSAIDs). XPF-001 does not have a rapid onset.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days